CLINICAL TRIAL: NCT04597840
Title: Multicenter, Prospective, Longitudinal and Randomized Comparison of Both the Clinical and Economic Impact of Biosynthetic Absorbable Mesh to the Surgical Standard of Care in Contaminated Incisional Hernia Repair
Brief Title: Biosynthetic Absorbable Mesh vs Standard of Repair for the Surgical Treatment of Infected Incisional Hernia
Acronym: COMpACT-BIO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69HCL20_0215
Record Dates: First submitted 2020-07-31; First posted 2020-10-22 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Ventral Hernia Repair
Keywords: ventral hernia repair; contaminated surgical field; infected incisional hernia; biosynthetic mesh

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The type of incisional hernia repair (simple suture or mesh reinforcement) will be masked to the primary outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biosynthetic mesh group (Experimental): Patient will undergo incisional hernia repair with biosynthetic mesh reinforcement. Based on the discretion of the surgeon, two types of biosynthetic mesh from different brand can be used: the Phasix mesh from BARD or the BioA mesh from GORE. These two biosynthetic meshes are resorbable, which means they are gradually absorbed by the body.
  Interventions: Procedure: Incisional hernia repair with reinforcement of biosynthetic mesh
- standard of repair group (Other): Patient will undergo incisional hernia repair according to the standard of repair, which is simple suture or mesh reinforcement (using synthetic or biological meshes).
  Interventions: Procedure: Incisional hernia repair with simple suture or synthetic mesh reinforcement.

INTERVENTIONS:
Procedure: Incisional hernia repair with reinforcement of biosynthetic mesh — The biosynthetic mesh (Phasix or Bio-A meshes) will be placed as a sublay in the retromuscular position to reinforce midline fascial closure. All the surgical procedure (including placement and fixation of the mesh) will be performed according to a standardized protocol.
  Arms: biosynthetic mesh group
Procedure: Incisional hernia repair with simple suture or synthetic mesh reinforcement. — Based on the discretion of the surgeon, the incisional hernia repair will be done by simple suture or by synthetic mesh reinforcement. All the surgical procedure (including placement and fixation of the mesh if applicable) will be performed according to a standardized protocol.
  Arms: standard of repair group

SUMMARY:
Incisional hernia is one of the most common complications of abdominal surgery and carries a significant burden for both patients and the economic health service. However, no consensus for the surgical treatment of incisional hernia in contaminated field is currently available. The purpose of the COMpACT-BIO study is to investigate the clinical and economic benefit of the use of biosynthetic mesh in contaminated incisional hernia repair.

DETAILED DESCRIPTION:
The current standard of incisional hernia repair is reinforcement with permanent synthetic mesh. However, permanent synthetic mesh is contraindicated in contaminated surgical field due to higher risk of postoperative infection. In order to resist to infection, absorbable meshes, such as biological and biosynthetic meshes, have been developped. However, some controversies exist about the clinical benefit of biological meshes in the long term. Reasons for theses controversies are their overall risk of complication and recurrence and the lack of consensus in which surgical technique to apply. Moreover, the financial cost of biological meshes is very high. Recently developed, biosynthetic meshes appear to be a promising option ; Compared to biological meshes, they seem to have several advantages. However, such data demonstrating the beneficial use of biosynthetic mesh in contaminated incisional hernia repair is not available. In this regard, the COMpACT-BIO study aims to investigate the clinical and economic benefit of the use of biosynthetic mesh in contaminated incisional hernia repair in comparison to the standard of repair. This is a multicenter, prospective, longitudinal and randomized study, which also offers a standardized technique of repair.

ELIGIBILITY:
All the following inclusion criteria must be fulfilled:

* Age ≥18 years old
* Physical status ASA < 4
* Patient with a mid-line IH
* Patient presenting with an IH without loss of domain
* Surgical indication in elective surgery
* "Potentially contaminated" grade III surgical environment according to the classification of the modified VHWG
* Cure of mid line IH feasible according to the defined standard technical modality (placement of a retromuscular prosthesis)
* No emergency surgical procedure
* Status of social insured or entitled to a social insurance
* Informed and signed consent of the patient after clear and appropriate information

The exclusion criteria are as follows:

* One or multiple incisional hernia out of the midline incision
* Pregnancy, breastfeeding, parturient or childbearing patients without contraception
* Known allergy to tetracyclines;
* Persons protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Rate of incisional hernia recurrence | 3 years after surgery
  The rate of incisional hernia recurrence will be evaluated by radiologic imaging.

SECONDARY OUTCOMES:
Days of hospitalization related to incisional hernia repair | For 3 years after surgery
  Number of days of hospitalization related to hernia repair-related complications will be reported.
Incidence of re-operation related to incisional hernia repair | For 3 years after surgery
  Incidence of incisional hernia repair-related complications leading to re-operation will be reported.
Incidence of wound events | 1 month from surgery date, then 3-, 6- 12-, 24- and 36 months from surgery date
  Incidence of incisional hernia repair-related wound complications, such as wound infection will be reported.
Incidence of revision surgery or interventional radiologic procedure | 1 month from surgery date, then 3-, 6- 12-, 24- and 36 months from surgery date
  Incidence of revision surgery or interventional radiologic procedure related incisional hernia repair-related wound complications will be reported.
Rate of early incisional hernia recurrence | 1 month from surgery date, then 3-, 6- 12-, 24- and 36 months from surgery date
  The rate of incisional hernia recurrence evaluated by physical examination and then confirmed by radiologic imaging will be reported.
Incisional hernia specific quality-of-life assessment | Pre and post-surgery (1 month from surgery date, then 3, 6, 12, 24 and 36 months from surgery date).
  Self reported clinical symptoms before and after incisional hernia repair will be done using a modified version of the Carolina Comfort Scale . Severity of pain and discomfort pre and post repair will be measured during different daily activities (item). Each item is scored 0-5 (0= no symptom ; 5= worst symptom).
Number of healing days | 1 month from surgery date, then 3-, 6- 12-, 24- and 36 months from surgery date
  At each clinical examination, the time between surgery and the end of median scar care will be measured.
Rate of screening failure | 48 months after the start of the study
  The proportion of patients who did not receive the surgical procedure proposed by the study, and the related reasons of screening failure will be reported.
Assessment of health care consumption related to health care status | pre and post-surgery (1 month from surgery date, then 3, 6, 12, 24 and 36 months from surgery date).
  The cost / quality ratio will be measured using the consumption of health care and the health status. In one hand, each health care action will be reported (by the patient or the caregiver) and then the total cost relative to the health care will be measured. In another hand, self-reported health status before and after incisional hernia repair will be done using the EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Passot G, Margier J, Kefleyesus A, Rousset P, Ortega-Deballon P, Renard Y, Bin S, Villeneuve L. Slowly absorbable mesh versus standard care in the management of contaminated midline incisional hernia (COMpACT-BIO): a multicentre randomised controlled phase III trial including a health economic evaluation. BMJ Open. 2022 Aug 25;12(8):e061184. doi: 10.1136/bmjopen-2022-061184. PMID 36008058